CLINICAL TRIAL: NCT05150028
Title: A Virtual Intervention to Improve Medication Adherence in Pediatric Cancer: MedSupport
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: I 2048021
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Medication Adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Pediatric parent/caregiver (Experimental): Questionnaires along with educational videos
  Interventions: Behavioral: Patient participation
- Clinicians (Experimental): Will complete pre and post survey about medication education practices
  Interventions: Other: Clinician barrier reports

INTERVENTIONS:
Behavioral: Patient participation — Questionnaire
  Arms: Intervention - Pediatric parent/caregiver
Other: Clinician barrier reports — How many times a 7 question Survey on medication education practices is opened
  Arms: Clinicians

SUMMARY:
To develop a cancer center level practice intervention to promote treatment adherence and reduce outcome disparities in pediatric cancer survivors

DETAILED DESCRIPTION:
To conduct a pilot study to assess the feasibility and acceptability of the Social Determinants of Adherence intervention

ELIGIBILITY:
Inclusion Criteria:

Parents/caregivers of pediatric patients must meet the following criteria to be eligible:

* Parents/guardians of child that has been diagnosed with any cancer.
* Parents/guardians of child with any cancer between age 0 and 18.
* Parents/guardians of child on home-based oral anti-cancer therapy or supportive care therapy.
* The clinician for the family agrees to participate in the study.

Exclusion Criteria:

* Participants will be excluded from this study if unwilling or unable to complete the assessment in English

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Retention rates | Up to 8 weeks
  Feasibility of intervention as assessed by retention rates

SECONDARY OUTCOMES:
Feasibility of universal SDOA screening | up to 8 weeks
  Will be assessed by results of SDOA questionnaire an 8 item questionnaire rated on a 5-point Likert scale (0-I never experienced this ; 5 - I experience this quite a lot)
Provider satisfaction with barrier reports | up to 8 weeks
  REDCap analytics will track the rate of opened barrier reports

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Bouchard, MD, Principal Investigator — Roswell Park Comprehensive Cancer Center
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States